CLINICAL TRIAL: NCT04527211
Title: Effectiveness and Safety of Ivermectin for the Prevention of Covid-19 Infection in Colombian Health Personnel at All Levels of Care, During the 2020 Pandemic: A Randomized Clinical Controled Trial
Brief Title: Effectiveness and Safety of Ivermectin for the Prevention of Covid-19 Infection in Colombian Health Personnel
Acronym: IveprofCovid19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Javeriana University (Other)
Responsible Party: Principal Investigator, Eduar d. Echeverri, MD Spec. and Clinical Epidemiologist, Javeriana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Epi1JaveCali
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Healthcare Worker Patient Transmission
Keywords: prophylaxis; ivermectin; COVID-19; health workers; SARS-CoV2
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: It will be performed a randomized, multicenter, triple-masked, placebo-controlled clinical experiment to determine the relative risk of SARS COV-2 infection, seroconversion, and clinically presenting disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Simple randomization will be done with a random number generator and masking will be maintained by concealing the allocation with opaque envelopes. The active medicine as the control will have the same presentation, color and taste, it will be differentiated by a pre-established code from the maker. This will maintain the concealment of patients, caregivers and evaluators. At the central level, only an intervention safety coordinator will know the assignment of each patient in case serious adverse events occur and the concealment needs to be lifted. The outcomes of interest will be obtained from the clinical history of the patients and through direct measurement in the follow-up visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Experimental): Oral administration of ivermectin 200 mcg/kg every week for seven weeks
  Interventions: Drug: Ivermectin
- Placebo (Placebo Comparator): Oral administration of placebo of similar characteristics every week for seven weeks
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — Oral administration of ivermectin 200 mcg/kg every week for seven weeks

SUMMARY:
It will be performed a randomized, multicenter, triple-masked, placebo-controlled clinical experiment to determine the effectiveness and safety of the administration to of ivermectin at a dose of 200 mcg/kg once a week for 7 weeks in a prophylactic treatment against SARS COV-2 infection in 550 Colombian health workers during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Introduction: In less than four months, an outbreak of severe pneumonia, initially identified in Wuhan (China), has spread to more than 185 countries and territories, leaving more than 1,835,000 people compromised and 113,362 deaths, according to statistics provided by Johns Hopkins University (1). Additionally, this outbreak has collapsed health systems in some countries and has begun to have a huge impact on the global economy.

The etiological agent, an RNA virus of the Coronaviridae family called SARS COV-2, is characterized by having a high contagion index (R0 = 1, 4 - 5, 5) (2), high virulence and lethality rates that can go up to 10% in some populations. The contagion of health workers has led to the loss of subjects with high social value to face the pandemic further weakening health systems. Because it is necessary to wait several months for the development, testing, approval and commercialization of a SARS COV-2 vaccine, there has been an urgent need to identify drugs that can offer a prophylactic effect for health workers who have high risk of being infected with the virus.

Recently, the in vitro antiviral effect of ivermectin was described to inhibit the invasive cellular action of SARS COV-2 (3), an effect explained by the HTA (Host Target Antivirals) model. Given the known safety and effectiveness of ivermectin in the treatment of parasitic infections in humans, this drug could be used prophylactically in health workers if the effects described on in-vitro studies are also present on in-vivo scenarios. However, so far, no study has shown the antiviral effects that ivermectin could have against SARS COV-2 or its effectiveness in reducing health complications caused by this virus in humans.

Objective: To determine the effectiveness and safety of the administration of ivermectin at a dose of 200 mcg/kg once a week for 7 weeks in a prophylactic treatment against SARS COV-2 infection in Colombian health workers during the COVID-19 pandemic.

Methods: It will be performed a randomized, multicenter, triple-masked, placebo-controlled clinical experiment to determine the relative risk of SARS COV-2 infection, seroconversion, and clinically presenting disease. In addition, the relative risk of requiring hospitalization or entering the intensive care unit was evaluated in doctors, nurses, respiratory therapists and assistants who have direct contact with patients with COVID-19. After being exposed to ivermectin prophylaxis or placebo for seven weeks, the results will be measured at eight weeks, with interim analyses to monitor the safety of the participating subjects.

Keywords: Coronavirus 2019, COVID-19, SARS-CoV2, ivermectin, prophylaxis, treatment, health workers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years old of any sex who work as health care workers, laboriously active during the recruitment of the study in health services that do not screen for the exclusion of acutely ill patients.
* Subjects who have not presented general symptoms such as general discomfort, fever, cough, dyspnoea or muscle pain in the last week.
* Subjects with negative COVID-19 serological antibody diagnostic tests.

Exclusion Criteria:

* Subjects considered as a resolved case of COVID-19 infection, according to guidelines from the Colombian National Institute of Health.
* Health personnel with social distancing due to close contact without personal protective equipment with confirmed patients of infection, or who are taking any medication as possible prophylaxis for COVID-19 (example; chloroquine, hydroxychloroquine, azithromycin)
* Health workers who have permits or temporary withdrawal from their hospital work for more than one week during the first month of the study.
* Subjects with known allergy to ivermectin.
* Women in a state of pregnancy or lactation.
* |Subjects with a body mass index less than 18.5 and greater than 35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-09-07 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-16 (Estimated)

PRIMARY OUTCOMES:
Clinical development of covid-19 disease during the intervention period | 8 weeks
  Development of of the disease according to the definitions of cases found in the guidelines from the Colombian National Institute of Health

SECONDARY OUTCOMES:
Seroconversion | 8 weeks
  Indicate if the patient had positive serological antibodies at the end of the study
Hospitalization requirement | 8 weeks
  Need for hospitalization independent of the level of complexity due to covid-19
Intensive Care Unit Requirement | 8 weeks
  ICU need due to Covid-19
Safety of the intervention | 8 weeks
  Adverse effect due to medication or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Eduar D. Echeverri, Dr., Principal Investigator — Pontificia Universidad Javeriana
Locations (1):
- Pontificia Universidad Javeriana, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No